CLINICAL TRIAL: NCT04796948
Title: A Phase I Study to Evaluate the Safety and Tolerability of Irinotecan Liposome in Combination With Oxaliplatin and 5-FU/LV in the Treatment of Advanced Pancreatic Cancer
Brief Title: A Study of Irinotecan Liposome in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-YLTKL-101
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Advanced Pancreatic Cancer

STUDY DESIGN:
Intervention Model Description: A dose-escalation and expansion study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan liposome；oxaliplatin；5-FU(Fluorouracil Injection)；LV(Calcium Folinate Injection) (Experimental): 1. irinotecan liposome: irinotecan liposome injection is irinotecan encapsulated in liposomes for i.v. infusion.
  2. oxaliplatin: oxaliplatin is a sterile, aqueous solution; 50mg/vial.
  3. 5-FU(Fluorouracil Injection): an aqueous, sterile, nonpyrogenic injectable solution available in 10ml/0.25g.
  4. LV(Calcium Folinate Injection): be supplied in vials containing 10ml/0.1g and available as an injectable solution.
  Interventions: Drug: Irinotecan liposome；oxaliplatin；5-FU(Fluorouracil Injection)；LV(Calcium Folinate Injection)

INTERVENTIONS:
Drug: Irinotecan liposome；oxaliplatin；5-FU(Fluorouracil Injection)；LV(Calcium Folinate Injection) — irinotecan liposome in combination with oxaliplatin and 5-FU/LV

SUMMARY:
To determine the safety and tolerability of irinotecan liposome in combination with oxaliplatin and 5-FU/LV in subjects with advanced pancreatic cancer who have not received prior systemic chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 70 years (including 18 and 70 years);
2. Patients with histologically or cytologically diagnosed pancreatic cancer (from pancreatic ductal epithelium), and clinical records show unresectable locally advanced or metastatic pancreatic cancer (stage III/IV based on the 8th Edition of the AJCC TNM staging for pancreatic cancer).
3. Have not received systemic anti-tumor therapy for the current stage of disease, including surgery (except stent placement), radiotherapy, chemotherapy, targeted therapy, immunotherapy or investigational therapy;
4. If the subject has previously received adjuvant chemotherapy, it is necessary to ensure that the time interval between the last dose and the first dose of this study is more than 12 months, and the adjuvant therapy-toxicity has recovered (judged as ≤ grade 1 based on CTCAE 5.0 criteria);
5. Must have at least one measurable lesion that can be taken as the target lesion (according to the RECIST v1.1 criteria);
6. Eastern Cooperative Oncology Group (ECOG) performance status score: 0 - 1 point;
7. Expected survival ≥3 months;
8. Major organs are functioning well

Exclusion Criteria:

1. Patients with pancreatic cancer originating from extrapancreatic ductal epithelium, including pancreatic neuroendocrine carcinoma, acinar cell carcinoma of the pancreas, pancreatoblastoma, and solid-pseudopapillary tumor;
2. Patients with known central nervous system metastases;
3. Patients carrying homozygous mutations of UGT1A1*28/*6 gene;
4. Severe gastrointestinal dysfunction;
5. Severe infection (> CTCAE grade 2), such as severe pneumonia, bacteremia, infection complications, etc. requiring inpatient treatment, occurred within four weeks before enrollment, and symptoms and signs of infection requiring intravenous antibiotic therapy (except for prophylactic antibiotics) occurred within two weeks before enrollment;
6. Received any of the following treatments:

1）Previously received treatment with irinotecan-containing regimens; 2）Received concomitant medications containing strong inhibitors/strong inducers of CYP3A4 or strong inhibitors of UGT1A1 within two weeks before enrollment; 3）Received the last anti-cancer treatment (including surgery, radiotherapy, etc.) within four weeks before enrollment; 4）Have received treatment with any other investigational drug/device within four weeks before enrollment; 5）Enrolled in another clinical study at the same time unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up.

7.Having experienced an arteriovenous thrombotic event, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism, within one year before enrollment; 8.Patients with cardiac clinical symptoms or diseases that are not well controlled, such as: (1) Patients with NYHA class 2 and above cardiac failure; (2) unstable angina; (3) myocardial infarction that occurred within one year; (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.

9.Patients who have suffered from malignant tumors other than pancreatic cancer before using the study drug for the first time, except those with low risk of metastasis and death (5-year survival rate >90%), such as adequately treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin; 10.Have any contraindication to either irinotecan liposome, irinotecan, 5-FU, calcium folinate, or oxaliplatin;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
MTD | 18 months
  Maximum tolerated dose for patients in combination treatment.
RP2D | 18 months
  Recommended phase II dose for patients in combination treatment.

SECONDARY OUTCOMES:
Frequency and severity of AEs/SAEs as Assessed by CTCAE v5.0 | From first dose to death; until the data cut off 18 months after the last subject is enrolled. The minimum time in follow up was 18 months.
  Through laboratory test, physical examination, vital signs,12-lead electrocardiogram (ECG), Echocardiogram, etc.;
Objective Response Rate (ORR) | From first dose to death; until the data cut off 18 months after the last subject is enrolled. The minimum time in follow up was 18 months.
  Number of reported responses (complete [CR] and partial [PR]) divided by the number of reported assessable patients.
Disease Control Rate (DCR) | From first dose to death; until the data cut off 18 months after the last subject is enrolled. The minimum time in follow up was 18 months
  Based on investigator reviewed radiographic tumour assessment and death.
Duration of Response (DoR) | From first dose to death; until the data cut off 18 months after the last subject is enrolled. The minimum time in follow up was 18 months.
  Based on investigator reviewed radiographic tumour assessment and death.
Progression-Free Survival (PFS) | From first dose to death; until the data cut off 18 months after the last subject is enrolled. The minimum time in follow up was 18 months.
  Based on change in tumour per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1
Overall Survival (OS) | From first dose to death; until the data cut off 18 months after the last subject is enrolled. The minimum time in follow up was 18 months.
  Based on investigator reviewed radiographic tumor assessment and death.
Cmax | 28days
  peak plasma concentration
Tmax | 28days
  time to peak concentration
AUC | 28days
  area under the plasma concentration versus time curve
t1/2z | 28days
  elimination half-life
Vss | 28days
  steady-state apparent volume of distribution
CL | 28days
  clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu Q, Zhao X, Wang X, Zhu R, Cheng Y, Xia T, Wu H, Tian H, Sun Y, Zhang M, Gao C, Fu D, Wu X, Zheng T, Yin X, Chen Y, Chen X, Li Z, Chen R, Yang X, Wang H, Wang Q, Han X, Wu W. Phase 1 trial of HR070803 (an Irinotecan liposome) in combination with 5-fluorouracil, leucovorin, and oxaliplatin for untreated advanced or metastatic pancreatic ductal adenocarcinoma. BMC Med. 2025 Jul 7;23(1):402. doi: 10.1186/s12916-025-04234-4. PMID 40619376